CLINICAL TRIAL: NCT05732272
Title: Improving Smoking Abstinence Outcomes in the African American Community Through Extended Treatment
Acronym: (KISV)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00148037
Record Dates: First submitted 2023-02-07; First posted 2023-02-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Treatment (Active Comparator): 250 participants will be randomly assigned to the standard treatment arm and receive 7 weeks of bupropion SR following standard dosing guidelines(150 mg once daily for 3 days, then 150mg twice daily for 7 weeks). Participants in this arm will also receive 8 smoking cessation counseling sessions consistent with the Clinical Practice Guidelines.
  Interventions: Drug: Bupropion
- Extended Treatment (Active Comparator): 250 participants will be randomly assigned to the extended treatment arm and receive 24 weeks of bupropion SR following standard dosing guidelines(150 mg once daily for 3 days, then 150mg twice daily for 24 weeks). Participants in this arm will also receive 8 smoking cessation counseling sessions consistent with the Clinical Practice Guidelines.
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Bupropion — 150 mg once daily for 3 days, then twice daily for the remainder of the treatment phase.

SUMMARY:
This study will evaluate the efficacy of extended bupropion(6 months) versus standard bupropion treatment (7 weeks) among African American daily smokers.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate extended use of bupropion with the goal of enhancing abstinence in African American daily smokers, including the full spectrum of light, moderate, and heavy smokers. A two-arm, randomized design will be used to evaluate the efficacy of extended (6 months) bupropion treatment compared to standard (7 weeks) bupropion treatment. Baseline randomization stratified by gender and cpd (≤10, >10cpd) will assign participants (N=500) to receive extended treatment (EXT; 24 weeks of bupropion, n=250) or standard treatment (ST; 7 weeks of bupropion, n=250). All participants will receive culturally-relevant, individualized smoking cessation counseling, including support for medication adherence, and will be followed through Month 12.

ELIGIBILITY:
Inclusion Criteria:

* African American
* age >18 years
* interested in quitting
* smoked >1 cpd for >1 years
* smoked on >25 days in the past month
* willing to take 6 months of study medication and complete all visits
* have a home address and functioning telephone number

Exclusion Criteria:

* Consistent with contraindications for bupropion:
* use of psychoactive medications
* history of alcohol or substance abuse within the past year
* binge drinking (>5 drinks on one occasion) >2 times in the past month
* history of seizures or head trauma; history of bulimia or anorexia nervosa
* pregnant (as measured by over the counter pregnancy test kit for women of child-bearing age only) or contemplating pregnancy; breast feeding
* myocardial infarction in the past 2 months
* reported use of opiates, cocaine, or stimulants
* unstable diabetes
* bupropion is a known inhibitor of the liver enzyme CYP2D6, so those taking drugs known to be higher metabolized by this enzyme (e.g., metoprolol, tamoxifen) will be excluded.
* use of stop smoking medications (bupropion, varenicline, nicotine replacement, fluoxetine, clonidine, buspirone, or doxepin) in the past 30 days
* planning to move from the Kansas City area in the next year
* other smoker in household enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Verified abstinence at Month 6 | Month 6
  Participants receiving extended bupropion treatment will have significantly higher Month 6 verified point-prevalence abstinence than participants receiving standard bupropion treatment.

SECONDARY OUTCOMES:
Adherence to medication | Week 4
  We will evaluate the concordance of a biological sample of bupropion level, observable pill count, and 3-day recall as measurements of medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Sanderson Cox, PhD, Principal Investigator — University of Kanas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No